CLINICAL TRIAL: NCT04105816
Title: Assessing the Reliability and Validity of Ultrasound to Evaluate Large Muscle Atrophy in the Lower Limbs
Brief Title: Ultrasound for Rectus Femoris Measurement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19 continually delayed in-person research
Sponsor: Robert Westermann (Other)
Responsible Party: Sponsor-Investigator, Robert Westermann, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201906778
Record Dates: First submitted 2019-09-22; First posted 2019-09-26 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Muscle Atrophy, Proximal; Muscle Atrophy; ACL Tear; Quadriceps Muscle Atrophy
Keywords: rectus femoris; ACL repair recovery; musculoskeletal ultrasound; quadriceps atrophy; validation
MeSH Terms: conditions — Muscular Atrophy; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adult Healthy Controls (Placebo Comparator): Subjects included in part I of this study will be healthy adult volunteers with no known musculoskeletal injury. Exclusion criteria will be those with identified musculoskeletal injury, non-English speaking persons, and women who are pregnant.
  Interventions: Device: 892.1550 Ultrasonic pulsed doppler imaging system; Diagnostic Test: Thigh circumference measurement
- Adult ACL Reconstruction Patients (Experimental): Subjects included in part II of the study will be adult volunteers undergoing anterior cruciate ligament reconstruction at the University of Iowa. Exclusion criteria will be non-English speaking persons, women who are pregnant, patients undergoing multi-ligament repair, patients undergoing ACL reconstruction revision, patients undergoing concomitant cartilage or meniscal repair procedures, and patients undergoing bilateral ACL reconstructions.
  Interventions: Device: 892.1550 Ultrasonic pulsed doppler imaging system; Diagnostic Test: Thigh circumference measurement

INTERVENTIONS:
Device: 892.1550 Ultrasonic pulsed doppler imaging system — Use of the ultrasound to measure quadriceps volume
Diagnostic Test: Thigh circumference measurement — Tape measure used to measure thigh circumference of all participating patients in the study at the same visit in which they receive ultrasound measurements of thigh muscles.

SUMMARY:
Postoperative protocols for orthopedic procedures on the lower limb often require a period of immobilization to protect the surgical site. The consequence of this immobilization is muscle atrophy which can be severe, delaying a patient's return to activity and predisposing them to recovery complications or subsequent injury (1)(2).

The current standard methods to assess lower limb muscle atrophy all have their respective limitations. Thigh circumference or isokinetic strength values are indirect measures of atrophy and can be inaccurate. Magnetic resonance imaging (MRI) of muscle cross-sectional area (CSA) is time-consuming and expensive. Computed tomography imaging of muscle CSA is expensive and exposes the patient to radiation (3). For these reasons, none of the current methods are ideal for regular use in the clinic.

Musculoskeletal ultrasound is a promising measurement tool to assess muscle atrophy in postoperative patients. Ultrasound is non-invasive, cost-effective, does not involve radiation, and can give direct images of muscle size (4). Musculoskeletal ultrasound requires further research on its potential as an evaluation tool for postoperative lower limb orthopedic patients-specifically, whether ultrasound is a reliable and valid tool for quadriceps size measurements.

DETAILED DESCRIPTION:
Lower limb surgeries, particularly knee surgeries, are prevalent procedures in US orthopedic departments. Many of these procedures require a postoperative period of immobilization, which may be lengthy for surgeries involving ligament reconstruction, fractures, meniscal repairs, or cartilage transplantation. This leg immobilization results in rapid and significant loss of skeletal muscle mass. Even for shorter periods of immobilization, atrophy occurs within as little as 5 days of immobilization in healthy subjects, and the largest extent of post-operative atrophy takes place during the first two weeks of being immobilized (1)(2).

Muscle atrophy can prolong recovery times and directly impact the safety of a patient's return to activity progression. Providers need a reliable, valid method of assessing postoperative muscle atrophy which is cost-effective, safe, and simple to implement in a clinical setting (4). The aim of this study is to demonstrate that ultrasounds are reliable and valid tools for measuring large lower limb stabilizers such as the rectus femoris. Upon proving reliability and validity, we aim to use the ultrasound to track and characterize rectus femoris atrophy after a common lower limb surgical procedure; anterior cruciate ligament (ACL) reconstruction. Success of this validation study would support the use of ultrasound to monitor large muscle atrophy after lower limb orthopedic surgical procedures, and to evaluate the impact of muscle health interventions. Our ultimate research aim is to develop a reliable, valid ultrasound measurement technique to evaluate promising perioperative interventions for attenuation of muscle atrophy following surgical procedures of the knee.

Patients and Methods:

Part I: Ultrasound measurements of the rectus femoris will be obtained in approximately 50 healthy volunteers. Thigh circumference measurements will be taken as well. The ultrasound (US) images will be de-identified with research identifier (ID) only and transferred from the US unit to a secured folder on a research drive, and associated only with basic demographic information such as age, gender, height, and weight. Ultrasounds currently in use at the UIHC Sports Medicine Clinic will be used. Measurements will be made at a point mid-way between the anterior superior iliac spine and the superior border of the patella.

Part II: Following validation in healthy controls, approximately 100 ACL reconstruction patients will be enrolled for a longitudinal study which utilizes the same ultrasound methods and equipment to track their rectus femoris size at a preoperative visit, and during the 6 week, 3 month, and 6 month standard postoperative follow-up visits. Thigh circumference measurements will be taken as well. The ultrasound images will be de-identified with research ID only and transferred from the US unit to a secured folder on a research drive, and associated only with basic demographic information such as age, gender, height, and weight; along with basic survey data on physical therapy adherence. The patients will not incur any cost from the ultrasound testing, and the ultrasound testing will occur at the same clinical location (UIHC Sports Medicine Clinic) as their follow-up visits.

Aim 1: Assess the inter-rater and intra-rater reliability of ultrasound for measuring skeletal size using a commercially available ultrasound unit.

Hypothesis 1: We hypothesize that ultrasound measures of rectus femoris will demonstrate both high intrarater and interrater reliability.

Aim 2: Assess the validity of ultrasound in measuring muscle size when utilized by a novice user as compared to a professional sonographer.

Hypothesis 2. The ultrasound will demonstrate high validity and ease of use when comparing novice and professionally obtained images.

Aim 3: Assess the accuracy of ultrasound in measuring muscle size compared to the literature standard measurement technique of thigh circumference.

Hypothesis 3: Ultrasound measurements will be equally or more accurate than thigh circumference measurements at detecting rectus femoris size differences between subjects, and ultrasound measurements will have less interrater and intrarater variability.

Aim 4: Develop a descriptive characterization of rectus femoris size parameters among a healthy young adult population.

Aim 5: Track and characterize rectus femoris atrophy in ACL reconstruction patients using the validated ultrasound methodology.

Hypothesis 4: Patients will show a statistically significant degree of rectus femoris atrophy between their preoperative visit measurement and their 6 week and 3 month follow up measurements.

Hypothesis 5: Patients will show a statistically significant degree of improvement in rectus femoris atrophy when comparing their 6 month visit measurements with their 6 week and 3 month visit measurements.

Hypothesis 6: There will not be a significant difference between the preoperative and 6 month postoperative rectus femoris measurements.

Hypothesis 7: Ultrasounds measurements will be equally or more sensitive at detecting significant rectus femoris atrophy in anterior cruciate ligament reconstruction (ACLR) patients compared to thigh circumference measurements.

Aim 6: Analyze how external factors impact rectus femoris atrophy in ACL reconstruction patients using the validated ultrasound methodology Hypothesis 8: Graft choice will impact rectus femoris atrophy and recovery. Hypothesis 9: Fewer physical therapy office visits will impact rectus femoris atrophy and recovery.

ELIGIBILITY:
Part 1 - Healthy Controls

Inclusion criteria will be:

Healthy adults with no known musculoskeletal injury

Exclusion criteria will be:

* Those with identified musculoskeletal injury
* Non-English speaking persons
* Women who are pregnant. Graduate medical education residents will be from the

Part 2 -

Inclusion criteria will be:

-Adult volunteers undergoing anterior cruciate ligament reconstruction at the University of Iowa

Exclusion criteria will be:

* non-English speaking persons
* women who are pregnant
* patients undergoing multi-ligament repair
* patients undergoing ACL reconstruction revision
* patients undergoing concomitant cartilage or meniscal repair procedure
* patients undergoing bilateral ACL reconstructions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity of musculoskeletal ultrasound use | 2 weeks
  Intra- and inter-rater validity compared to thigh circumference measurements. For inter-rater, intra-rater , and the comparison between professional and novice users, for muscle cross sectional area/thickness, we will use inter-rater correlation coefficient (ICC), kappa statistic, and Bland-Altman plot analysis. These analyses will help us determine validity of the ultrasound measuring device. Measurements of the contralateral limb will be used as internal controls. Due to the nature of this study, a power analysis is not needed, since it is a validity/characterization study and we are not looking to find a specific difference between the two types of users.
Reliability of musculoskeletal ultrasound use | 2 weeks
  Intra- and inter-rater reliability, reliability compared to thigh circumference measurements. For inter-rater, intra-rater reliability, and the comparison between professional and novice users, for muscle cross sectional area/thickness, we will use inter-rater correlation coefficient (ICC), kappa statistic, and Bland-Altman plot analysis. These analyses will help us determine reliability of the ultrasound measuring device and the measuring technique between individual users and between measurements by the same individual. Measurements of the contralateral limb will be used as internal controls. Due to the nature of this study, a power analysis is not needed, since it is a validity/characterization study and we are not looking to find a specific difference between the two types of users.
Amount of quadriceps atrophy using musculoskeletal ultrasound following anterior cruciate ligament reconstruction | 6 months
  Change in the operative leg versus non-operative leg muscle cross sectional area/thickness will be determined. The degree of change in the operative leg versus the non-operative leg will be evaluated for significant differences. The total number of patients with significant differences between their operative and non-operative legs will be recorded for each time point in the study. The mean and median amount of change at each time point in the operative leg versus the non-operative leg will constitute the "amount of quadriceps atrophy" outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Westermann, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Sports Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No